CLINICAL TRIAL: NCT06258954
Title: Effect of 3D-printed Reconstruction Automated Matching System in Selecting the Size of Left Double-lumen Tube
Brief Title: Effect of 3D-printed Reconstruction System in Size of Left DLT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yihao Zhu, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: scchec-20240128
Record Dates: First submitted 2024-01-28; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Cancer of Lung; Lung Isolation
Keywords: Lung isolation; double-lumen tube; Three-dimensional reconstruction
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D group (Experimental): Using automatic comparison software for 3D reconstruction to determine the size of DLT.
  Interventions: Other: 3D reconstruction
- control group (Placebo Comparator): The size of DLT is based on patient's sex and height.
  Interventions: Other: traditional method for selecting double lumen tube

INTERVENTIONS:
Other: 3D reconstruction — 3D reconstruction based on CT data and It reconstructs the trachea and bronchus and compares them with the DLT, predicting the most suitable size of the DLT for lung isolation.
  Arms: 3D group
Other: traditional method for selecting double lumen tube — In control group, the size of DLT is based on patient's sex and height.
  Arms: control group

SUMMARY:
The precise and accurate size of DLT is a prerequisite to ensure its accurate position of its placement. Three-dimensional (3D) reconstruction technology can accurately reproduce the tracheobronchial structure to improve the correct size selection of DLT. To make it simpler, the investigators developed an automatic comparison software for 3D reconstruction based on computed tomography data (3DRACS). In this study, the investigators aimed to prove that 3DRACS is much more efficient in endobronchial intubation compared to the traditional method.

DETAILED DESCRIPTION:
Lung isolation techniques are commonly used to facilitate surgical exposure and to provide single-lung ventilation for patients undergoing various intra-thoracic procedures. Lung isolation is primarily accomplished with a double-lumen tube (DLT) or bronchial blocker. One published study showed that residents with limited experience had a 40% error rate in accurately placing a DLT. The accurate choice of the size of DLT is a prerequisite for good lung isolation.Currently, There is lack of proper objective criteria for selecting size of DLT. DLT size selection is estimated empirically using the patient's height and sex, and studies have shown that the size of DLT according CT images of the chest is more accurate than experience. The investigators have developed an automatic comparison software for 3D reconstruction based on CT data (3DRACS). It reconstructs the trachea and bronchus and compares them with the DLT, predicting the most suitable size of the DLT for lung isolation. The aim of this study was to compare whether the use of 3DRACS to select a DLT size compared to conventional empirical selection methods could improve incidence of DLT intubation success and reduce airway injury.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. American Society of Anesthesiologists Physical Status (ASA-PS) I-III.
3. Planned to receive lung resection surgery during lung isolation techniques by using DLT.
4. Signed informed written consent.

Exclusion Criteria:

The participant experiences any of the following：

1. Spinal malformation,
2. Expected difficult airway
3. Tracheal stenosis
4. Tracheal tumor
5. Bronchial tumor
6. Distorted airway anatomy
7. Tumors of the mouth or neck

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
the success rates of placement of left DLT without FOB | After intubation，an average of 2 hours
  Conventional blindly endobronchial intubation is performed firstly and clinical verification was made by the same anesthesiologist, followed by the supervising anesthesiologist using a FOB to check DLT position and successful intubation was considered if the position was proper.

SECONDARY OUTCOMES:
The time of completing the left DLT's position | After intubation，an average of 2 hours
  There are two different situations that we need to describe. First, it starts from the cuff of left DLT crosses the vocal cords, and stops when the left DLT position succeeds without FOB(attempts≤3）. A stopwatch is used for this purpose, where it is ON when the cuff of left DLT crosses the vocal cords and stops when intubating anesthesiologist considers the left DLT is correctly positioned. Second, it starts from the cuff of left DLT crosses the vocal cords and stops when positioning successfully with FOB after three attempts all fail. Each attempt is defined as returning the bronchial lumen of the left DLT to the trachea and then attempting to reinsert it.
The number of the patients who need to change the size of the left DLT | After intubation，an average of 2 hours
  If the position of the left DLT under the FOB guidance doesn't match and the intubation fails because of the improper size of the left DLT, we need to change another left DLT.
Appropriate standard for the left DLT | After intubation，an average of 2 hours
  Objective criteria is injecting air into the cuff. When the pressure inside the left DLT is 25 mmHg, it will be stopped and connected to the anesthesia machine. And the air leakage phenomenon is adjusted when the peak pressure is lower than 30 cm H2O. Oversized left DLT is defined that good pulmonary isolation could be achieved by injecting <1 ml of air into the bronchial cuff and <2 ml of air into the main tracheal cuff, while more than 3 or 6 ml of air into the two cuff is defined undersized left DLT.
Lung collapse | At 10 and 20 minute after pleurotomy
  Ten and 20 min after pleurotomy, the degree of pulmonary atrophy is assessed by a chest surgeon unaware of the grouping with an eleven-point Likert scale with 0 marked as no pulmonary atrophy at all and 10 as most perfect lung collapse.
Grading of the airway injury | After extubation，an average of 1 hours
  it will be done by a trained anesthesiologist with over 10 years of FOB experience, The severity of the tracheal injury is defined as mild (redness, edema, one to three speckled hemorrhagic lesions), moderate (over 3 mild lesions or one diffuse hemorrhagic lesion), and severe (more than 2 diffuse hemorrhagic lesions) The type of lesions in vocal cords is classified into edema with inflamed mucosa, petechiae (small red spots on the mucosa), and hematoma (bleeding into the mucosa).
Postoperative sore throat and hoarseness | 1, 2 days after surgery
  they are defined as persistent resting pain in the throat region, where throat pain scores are assessed using VAS score i.e., 0 for no pain, and 10 for unbearable pain, while hoarseness is defined as a change in the quality of voice observed by the patient.
Oxygenation during one-lung ventilation | At the end of surgery.
  it is defined as the area under the curve of the SpO2/FiO2 ratio during OLV. The SpO2 and FiO2 values are automatically collected by the monitor at 30-second intervals and any abnormal data due to equipment or human error is replaced with the previous correct data.
Times of using FOB | At the end of surgery.
  The times of using FOB guiding to place the left DLT correctly after three attempts all fail.

CONTACTS AND LOCATIONS:
Overall Officials: Yihao Zhu, master, Principal Investigator — department of anesthesiology, sichuan cancer hospital

IPD SHARING:
Plan to Share IPD: No
Data are available on reasonable request. The raw data are available from the corresponding author with applicable reason after publishing findings to a peer-reviewed journal.

REFERENCES:
- [Derived] Li L, Zhu Y, Yin F, Yu H, Wang H, Xu Y, Fei F, Liu W, Duan B, Wang F, Jia Y, Zhang H. Effect of a 3D-printed reconstruction automated matching system for selecting the size of a left double-lumen tube: a study protocol for a prospective randomised controlled trial. BMJ Open. 2024 May 15;14(5):e085503. doi: 10.1136/bmjopen-2024-085503. PMID 38754878